CLINICAL TRIAL: NCT05244369
Title: Efficacy of Acupuncture in Patients With Lower Extremity Amputation With Neuroma: A Prospective Randomized Controlled Study
Brief Title: Efficacy of Acupuncture in Patients With Lower Extremity Amputation With Neuroma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Specialist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2021-06

CONDITIONS: Neuroma Amputation
Keywords: Lower Extremity Amputation with Neuroma; Acupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture+TENS group (Active Comparator): Acupuncture application twice a week - a total of 8 sessions, and rehabilitation program consisting of joint range of motion, stretching and strengthening exercises for 30 minutes for 5 days a week for 4 weeks, current frequency 60-100 Hz to stump tip, impulse duration 100 microseconds transcutaneous electrical nerve stimulation (TENS) will be applied.
  Interventions: Procedure: Acupuncture+TENS
- Only TENS group (Other): A rehabilitation program consisting of joint range of motion, stretching, and strengthening exercises for 30 minutes, 5 days a week for only 4 weeks, and transcutaneous electrical nerve stimulation (TENS) with a current frequency of 60-100 Hz and an impulse duration of 100 microseconds will be applied.
  Interventions: Other: Only TENS

INTERVENTIONS:
Other: Only TENS — Rehabilitation program consisting of joint range of motion, stretching and strengthening exercises for 30 minutes, 5 days a week for only 4 weeks, and application of transcutaneous electrical nerve stimulation (TENS) to the tip of the stump
  Arms: Only TENS group
Procedure: Acupuncture+TENS — acupuncture application twice a week - a total of 8 sessions, rehabilitation program consisting of exercises 5 days a week for 4 weeks and transcutaneous electrical nerve stimulation (TENS) to the stump tip.
  Arms: Acupuncture+TENS group

SUMMARY:
Neuroma often occurs after major nerve damage or transection and can be diagnosed with pain at the tip of the stump, positive tinel, imaging (USG/MR). Various treatment methods are used for neuropathic pain, including pharmacological agents, intralesional steroid and local anesthetic injection, alcohol, phenol, radiofrequency or cryotherapy, ablation and surgical applications. Exercise (ROM and relaxation), TENS, biofeedback, hypnosis, acupuncture, psychotherapy, mirror therapy can be used in the treatment of neuropathic pain in amputees. In this study, the investigators aimed to examine the effectiveness of acupuncture on pain, neuroma size and functional status in individuals with lower extremity amputation with neuroma.

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, controlled trial. Thirty six people who met the inclusion criteria will randomized into two groups of 18 people. The first group will be designated as acupuncture therapy group and patients in the second group will be designated as the control group. Patients will be evaluated with visuel analog scale (10cm-VAS), LANSS (Self-Leeds Assessment of Neuropathic Symptoms and Sign) scale, Locomotor Capacity Index, 2-minute walking test, USG measurement. The patients will be evaluated at the beginning of the treatment (0.month), the end of the treatment (1st month), and the 4th month.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Having a diagnosis of lower extremity amputation
* Consent to be included in the study
* Having a complaint of pain

Exclusion Criteria:

Exclusion Criteria for the Acupuncture+TENS group

* Conditions in which acupuncture is strictly contraindicated (inflamed, infected or impaired skin, spontaneous bleeding, metal allergy, fear of needles, unstable diabetes mellitus patients, history of unstable epilepsy or unexplained convulsions, unstable acute cardiac arrhythmia or heart failure , heart valve disease or history of replacement surgery, presence of lymphedema)
* Lack of consent to be included in the study
* There are situations where TENS application is inconvenient

Exclusion Criteria for only TENS group

* There are situations where TENS application is inconvenient
* Lack of consent to be included in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
LANSS (Self-Leeds Assessment of Neuropathic Symptoms and Sign) | baseline, change from baseline VAS at 4 and 16 weeks
  The LANSS scale consists of two parts. If the score is 12 and above, it will be classified as neuropathic, and if it is below 12, it will be classified as nociceptive pain
Locomotor Capacity Index | baseline, change from baseline VAS at 4 and 16 weeks
  the patient's ability to perform 14 activities with the prosthesis will be evaluated. The total maximum score is 42, and the higher the total score, the higher the locomotor capacity.
10-point VAS | baseline, change from baseline VAS at 4 and 16 weeks
  The overall prosthesis satisfaction and socket comfort of the patients will be evaluated with a 10-point VAS. Patients will be asked to rate their condition from 0 (none) to 10 (maximum).
2-minute walking test | baseline, change from baseline VAS at 4 and 16 weeks
  the distance he walked at the end of two minutes will be recorded in meters (m).
ultrasonographic measurement | baseline, change from baseline VAS at 4 and 16 weeks
  The size of the neuroma will be visualized with a 7.5-12 MHz linear transducer (LOGIQ 7 Pro; GE Yokogawa medical system, Tokyo, Japan) USG and measured by the same clinician

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özcan, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No